CLINICAL TRIAL: NCT03841435
Title: Feasibility Study of Hypofractionated Radiotherapy in the Setting of Recurrent Diffuse Intrinsic Pontine Glioma
Brief Title: Hypofractionated Radiotherapy for Recurrent DIPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Luke Pater, Associate Professor of Radiation Oncology, Mediacal Director, West Chester Hospital Radiotherapy, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-2183
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Radiotherapy (Experimental): 15 Gy given in 3 fractions over 2 weeks
  Interventions: Radiation: Hypofractionated Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated Radiotherapy — Radiotherapy Treatment, totaling 15 Gy, will be given in 3 fractions over 2 weeks.

SUMMARY:
This study evaluates the feasibility of hypofractionated radiotherapy (RT) in the palliative treatment of recurrent diffuse intrinsic pontine glioma (DIPG). Participants will receive 15 Gy in 3 fractions as opposed to the standard 20 Gy in 10 fractions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≤30 years of age
2. Patients must have a diagnosis of progressive DIPG.
3. Received prior IMRT based definitive radiotherapy to a dose of ≥54 Gy.
4. The patient and or parent/legal guardian must be physically and mentally capable of signing the consent form of their own volition.
5. Steroids dosage must be unchanged for 5 days.
6. No Bevacizumab within 21 days (Half-life 11 days ~)

Exclusion Criteria:

1. Patients with incomplete medical records
2. Patients with prior history of reirradiation for DIPG
3. Life expectancy < or equal to 1 month
4. Pregnant women
5. Age >30
6. Prisoners
7. Concurrent systemic therapy at the time of reirradiation
8. Physically or mentally incapable of signing the consent form of their own volition
9. < 6 mos time interval between completion of initial RT to start of reRT.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Post Radiation Toxicity | Through Study Completion, an average of 1 year
  RTOG common toxicity criteria grade 0-5

SECONDARY OUTCOMES:
Change in Quality of Life score | Pre-RT, 2 weeks, 1 month, 3 months and every 3 months there-after post RT
  Patient reported quality of life via Pediatric Quality of Life Inventory Version 4.0
Radiographic Response | 1 month
  Physician documented change of tumor from pre-RT MRI as compared to 1 month post-RT MRI
Progression Free Survival | Through Study Completion, an average of 1 year
  Time to clinical, symptomatic or radiographic evidence of disease progression
Overall Survival | Through Study Completion, an average of 1 year
  Time to patient death
Steroid Requirement | Through Study Completion, an average of 1 year
  Use of steroids post-RT

CONTACTS AND LOCATIONS:
Overall Officials: Luke E Pater, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be kept confidential and will not be shared with other researchers

REFERENCES:
- [Background] Ostrom QT, Gittleman H, Farah P, Ondracek A, Chen Y, Wolinsky Y, Stroup NE, Kruchko C, Barnholtz-Sloan JS. CBTRUS statistical report: Primary brain and central nervous system tumors diagnosed in the United States in 2006-2010. Neuro Oncol. 2013 Nov;15 Suppl 2(Suppl 2):ii1-56. doi: 10.1093/neuonc/not151. No abstract available. PMID 24137015
- [Background] Vanan MI, Eisenstat DD. DIPG in Children - What Can We Learn from the Past? Front Oncol. 2015 Oct 21;5:237. doi: 10.3389/fonc.2015.00237. eCollection 2015. PMID 26557503
- [Background] Fangusaro J. Pediatric high-grade gliomas and diffuse intrinsic pontine gliomas. J Child Neurol. 2009 Nov;24(11):1409-17. doi: 10.1177/0883073809338960. Epub 2009 Jul 28. PMID 19638636
- [Background] Fontanilla HP, Pinnix CC, Ketonen LM, Woo SY, Vats TS, Rytting ME, Wolff JE, Mahajan A. Palliative reirradiation for progressive diffuse intrinsic pontine glioma. Am J Clin Oncol. 2012 Feb;35(1):51-7. doi: 10.1097/COC.0b013e318201a2b7. PMID 21297433
- [Background] Merchant TE, Boop FA, Kun LE, Sanford RA. A retrospective study of surgery and reirradiation for recurrent ependymoma. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):87-97. doi: 10.1016/j.ijrobp.2007.09.037. PMID 18406885
- [Background] Liu AK, Foreman NK, Gaspar LE, Trinidad E, Handler MH. Maximally safe resection followed by hypofractionated re-irradiation for locally recurrent ependymoma in children. Pediatr Blood Cancer. 2009 Jul;52(7):804-7. doi: 10.1002/pbc.21982. PMID 19260098
- [Background] Bouffet E, Hawkins CE, Ballourah W, Taylor MD, Bartels UK, Schoenhoff N, Tsangaris E, Huang A, Kulkarni A, Mabbot DJ, Laperriere N, Tabori U. Survival benefit for pediatric patients with recurrent ependymoma treated with reirradiation. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):1541-8. doi: 10.1016/j.ijrobp.2011.10.039. Epub 2012 Jan 13. PMID 22245198
- [Background] Iqbal MS, Lewis J. An overview of the management of adult ependymomas with emphasis on relapsed disease. Clin Oncol (R Coll Radiol). 2013 Dec;25(12):726-33. doi: 10.1016/j.clon.2013.07.009. Epub 2013 Aug 20. PMID 23972764
- [Background] Mayer R, Sminia P. Reirradiation tolerance of the human brain. Int J Radiat Oncol Biol Phys. 2008 Apr 1;70(5):1350-60. doi: 10.1016/j.ijrobp.2007.08.015. Epub 2007 Nov 26. PMID 18037587
- [Background] Massimino M, Biassoni V, Miceli R, Schiavello E, Warmuth-Metz M, Modena P, Casanova M, Pecori E, Giangaspero F, Antonelli M, Buttarelli FR, Potepan P, Pollo B, Nunziata R, Spreafico F, Podda M, Anichini A, Clerici CA, Sardi I, De Cecco L, Bode U, Bach F, Gandola L. Results of nimotuzumab and vinorelbine, radiation and re-irradiation for diffuse pontine glioma in childhood. J Neurooncol. 2014 Jun;118(2):305-312. doi: 10.1007/s11060-014-1428-z. Epub 2014 Apr 3. PMID 24696052
- [Background] Lassaletta A, Bartels U, Strother D, et al. Hg-57re-irradiation in patients with diffuse intrinsic pontine gliomas, an update on the canadian experience. Neuro-Oncology 2016;18:iii60-iii61.
- [Background] Freese C, Takiar V, Fouladi M, DeWire M, Breneman J, Pater L. Radiation and subsequent reirradiation outcomes in the treatment of diffuse intrinsic pontine glioma and a systematic review of the reirradiation literature. Pract Radiat Oncol. 2017 Mar-Apr;7(2):86-92. doi: 10.1016/j.prro.2016.11.005. Epub 2016 Nov 23. PMID 28274399
- [Background] Hoffman LM, Plimpton SR, Foreman NK, Stence NV, Hankinson TC, Handler MH, Hemenway MS, Vibhakar R, Liu AK. Fractionated stereotactic radiosurgery for recurrent ependymoma in children. J Neurooncol. 2014 Jan;116(1):107-11. doi: 10.1007/s11060-013-1259-3. PMID 24078173
- [Background] Mayo C, Yorke E, Merchant TE. Radiation associated brainstem injury. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S36-41. doi: 10.1016/j.ijrobp.2009.08.078. PMID 20171516
- [Background] Freeman CR, Krischer JP, Sanford RA, Cohen ME, Burger PC, del Carpio R, Halperin EC, Munoz L, Friedman HS, Kun LE. Final results of a study of escalating doses of hyperfractionated radiotherapy in brain stem tumors in children: a Pediatric Oncology Group study. Int J Radiat Oncol Biol Phys. 1993 Sep 30;27(2):197-206. doi: 10.1016/0360-3016(93)90228-n. PMID 8407392
- [Background] Packer RJ, Boyett JM, Zimmerman RA, Rorke LB, Kaplan AM, Albright AL, Selch MT, Finlay JL, Hammond GD, Wara WM. Hyperfractionated radiation therapy (72 Gy) for children with brain stem gliomas. A Childrens Cancer Group Phase I/II Trial. Cancer. 1993 Aug 15;72(4):1414-21. doi: 10.1002/1097-0142(19930815)72:43.0.co;2-c. PMID 8339232
- [Background] Packer RJ, Boyett JM, Zimmerman RA, Albright AL, Kaplan AM, Rorke LB, Selch MT, Cherlow JM, Finlay JL, Wara WM. Outcome of children with brain stem gliomas after treatment with 7800 cGy of hyperfractionated radiotherapy. A Childrens Cancer Group Phase I/II Trial. Cancer. 1994 Sep 15;74(6):1827-34. doi: 10.1002/1097-0142(19940915)74:63.0.co;2-q. PMID 8082086